CLINICAL TRIAL: NCT03290079
Title: Phase II Study of Pembrolizumab and Lenvatinib in Advanced Well-differentiated Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19207
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Carcinoma; Neuroendocrine Cancer
Keywords: well-differentiated neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: Simon 2-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab & Lenvatinib treatment (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks, in addition to 20 mg Lenvatinib by mouth every day of each 3 week cycle. Estimated average length of treatment per participant: 4 months.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg Pembrolizumab by IV on Day 1 of each 3 week cycle.
  Other Names: Keytruda®
Drug: Lenvatinib — 20 mg Lenvatinib by mouth every day of each 3 week cycle
  Other Names: Lenvima®

SUMMARY:
The purpose of this study is to:

* Assess overall radiographic response rate (ORR)
* Assess progression-free survival (PFS)
* Test the safety and tolerability of Pembrolizumab in combination with lenvatinib

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis/Condition for entry into the trial: Metastatic well differentiated neuroendocrine tumors of primary lung, thymic, small bowel and colorectal origin (including unknown primary)
* Evidence of radiographic disease progression with scan documenting progression occurring within 8 months of signing informed consent
* At least two prior lines of systemic treatment. If the only prior line of treatment was adjuvant or neoadjuvant, patient must have completed treatment within 12 months. There is no limit to number of prior therapies.
* Willing and able to provide written informed consent/assent for the trial.
* ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function and laboratory values. All screening labs should be performed within 14 days of treatment initiation.
* Females of childbearing potential (FOCBP) should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication.
* FOCBP must agree to use adequate contraception as outlined in study documentation for the course of the through 120 days after the last dose of study medication.
* Male participants of childbearing potential must agree to use an adequate method of contraception as outlined in study documentation, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Poorly differentiated neuroendocrine carcinoma
* Pancreatic neuroendocrine tumor
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* A diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Potential participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If have received major surgery within 3 weeks, must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility.
* Serious non-healing wound, ulcer or bone fracture
* Has pre-existing >/= Grade 3 gastrointestinal (GI) or non-GI fistula
* Has significant cardiovascular impairment within 12 months of the first dose of study drug
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Potential participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* An active infection requiring systemic therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has received prior therapy with a tyrosine kinase inhibitor (TKI) (e.g.; sunitinib, pazopanib, cabozantinib)
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg, despite optimal medical management
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic, attacks, DVT within the past 6 months
* Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR) monitoring.(Treatment with low molecular weight heparin (LMWH) is allowed)
* Marked baseline prolongation of QT/QTc interval (QTc interval ≥ 480 msec) using the Fridericia method (QTc = QT/RR0.33) for QTc analysis
* Clinically significant bleeding within 4 weeks
* Medical need for the continued use of potent inhibitors/inducers of CYP3A4
* Creatinine clearance <30 mL/min
* Any condition that impairs patient's ability to swallow whole pills or gastrointestinal malabsorption that, in the investigator's opinion, might affect absorption of lenvatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab & Lenvatinib Treatment
Started | 20
Completed | 18
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab & Lenvatinib Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Radiographic Response Rate (ORR)
Description: Response Evaluation Criteria in Solid Tumors (RECIST) based response rate. Complete Response (CR): Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (SLD) of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest). The SLD must also demonstrate an absolute increase of at least 5mm. (Two lesions increasing from 2 mm to 3 mm, for example, does not qualify). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 12 months
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab & Lenvatinib Treatment
Number analyzed (Participants) | 18
proportion of participants | .1 [.03 to .30]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR, defined as the time from first documented evidence of Complete Response (CR) or Partial Response (PR) until disease progression or death due to any cause, whichever occurs first.
Time Frame: Up to 12 months
Population: Evaluable participants
Measure: Mean (Full Range); unit: months
Arm/Group | Pembrolizumab & Lenvatinib Treatment
Number analyzed (Participants) | 18
months | 6.5 [4.8 to 7.4]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, defined as the time from initial treatment to the first documented disease progression according to RECIST 1.1, or death due to any cause, whichever occurs first.
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab & Lenvatinib Treatment
Number analyzed (Participants) | 20
months | 8 [5.8 to 10.2]

4. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from initial treatment until death from any cause.
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab & Lenvatinib Treatment
Number analyzed (Participants) | 20
percentage of participants | 70 [48.1 to 84.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment to 30 days after cessation of treatment, an average of 8.5 months. Patients were followed for survival only for 12 months.
Arm/Group | Pembrolizumab & Lenvatinib Treatment
All-Cause Mortality (participants affected / at risk) | 6/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab & Lenvatinib Treatment (N=20)
Kidney Infection (Infections and infestations) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Disease Progression (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) — COVID-19
Infections and infestations - Other (Infections and infestations) | 1 (1) — human metapneumovirus
Hypotension (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Death, NOS (General disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hip pain (General disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab & Lenvatinib Treatment (N=20)
Abdominal Pain (Gastrointestinal disorders) | 11 (18)
Diarrhea (Gastrointestinal disorders) | 11 (15)
Constipation (Gastrointestinal disorders) | 7 (10)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 4 (6)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — mucus in stool
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — hernia
Belching (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 12 (24)
Fever (General disorders) | 5 (6)
Pain (General disorders) | 5 (6)
Edema limbs (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (4)
Flu like symptoms (General disorders) | 2 (2)
Facial pain (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (13)
Dizziness (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (4)
Lethargy (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 15 (27)
Hypotension (Vascular disorders) | 5 (6)
Flushing (Vascular disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (9)
Pericardial effusion (Cardiac disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Weight loss (Investigations) | 8 (12)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Thyroid stimulating hormone increased (Investigations) | 3 (3)
Electrocardiogram T wave abnormal (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Investigations - Other (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 8 (12)
Hematuria (Renal and urinary disorders) | 1 (3)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 6 (6)
Endocrine disorders - Other (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 3 (4)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (2)
Eye disorders - Other (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT03290079/Prot_SAP_000.pdf